CLINICAL TRIAL: NCT01058187
Title: Assessment of Fatty Acids in Infants' Blood Cells When Consuming Infant Formula Containing Long-Chain Polyunsaturated Fatty Acids
Status: Completed | Type: Observational
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: University of Alberta (Other)
Responsible Party: Deolinda Scalabrin, M.D., Mead Johnson Nutrition
Other Study IDs: 6000
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Levels of Fatty Acids in the Blood Cells of Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Control: Marketed cow milk-based infant formula containing DHA and ARA
- Investigational 1: Cow milk-based infant formula with differing level of ARA from Control formula
- Investigational 2: Cow milk-based infant formula with a differing level of ARA from Control

SUMMARY:
To compare amounts of DHA, ARA, and other fatty acids in the blood cells of infants consuming infant formulas containing differing levels of fatty acids

ELIGIBILITY:
Inclusion Criteria:

* Singleton birth
* 12-25 days of age
* Gestational age of 37-42 weeks
* Solely formula fed for at least 24 hours prior to randomization
* Birth weight 2500 g - 4000 g

Exclusion Criteria:

* Serious concurrent illness or congenital malformation
* Systemic or congenital infection
* Immunocompromised
* History of intolerance or allergy to cow milk
* Maternal autoimmune disorder
* Participation in another clinical study

Ages: 12 Days to 25 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants 12-25 days of age
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Clandinin, Ph.D., Principal Investigator — University of Alberta
Locations (1):
- Alberta Institute for Human Nutrition, University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Miklavcic JJ, Larsen BM, Mazurak VC, Scalabrin DM, MacDonald IM, Shoemaker GK, Casey L, Van Aerde JE, Clandinin MT. Reduction of Arachidonate Is Associated With Increase in B-Cell Activation Marker in Infants: A Randomized Trial. J Pediatr Gastroenterol Nutr. 2017 Mar;64(3):446-453. doi: 10.1097/MPG.0000000000001283. PMID 27276431